CLINICAL TRIAL: NCT06139900
Title: The Effect of Different Visual Stimuli Provided by Virtual Reality on Postural Control in Healthy Subject
Brief Title: How Virtual Reality is Impacting Balance: An Examination of Postural Stability
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: 202106077
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: balance; postural control; virtual reality; visual
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment — No intervention will be applied to the participants. Postural stability will be evaluated in the virtual reality environment and real environment.

SUMMARY:
There are several studies examining the effects of different sensory stimuli on balance in healthy young people. Our study will especially explain how the same environment will affect postural control, when projected into VR environment. In this way, we aim to contribute to the literature and virtual reality programs used in rehabilitation.

DETAILED DESCRIPTION:
Thanks to the development of technology in recent years, virtual reality applications have started to be included in physiotherapy. Virtual reality is used in both clinical and academic studies for the purpose of training rather than evaluation. In the literature, it has been emphasized that traditional balance training does not have any superiority over virtual reality and virtual reality training can be used as a practical alternative in the long term (12,13). Furthermore, the feedback provided by virtual reality games is effective in the patient's participation in the treatment. Different visual stimuli created using virtual reality can affect postural control in different ways (14). In addition, there is no study comparing the effect of real image and virtual reality image on postural control by transferring the current environment to virtual reality. The aim of this study is to reflect the real environment to virtual reality; To explain how postural control is affected by eyes closed, eyes open and in virtual reality. Two hypotheses were determined in this study.

H0: There is no significant difference between the real environment and three virtual environment on postural control in healhty subject.

H1: There is a significant difference between the real environment and three virtual environment on postural control in healthy subject.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30
* The absence of any medical diagnosis
* Having visual acurity or corrected visual acurity
* Being volunteer

Exclusion Criteria:

* The presence of any medical diagnosis
* The presence of any neurologic symptoms
* The presence of any sensory problems
* The presence of any balance problems
* The presence of any vestibular problems
* Previous ortophedic surgery
* The use of an additional assistive device

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Voluntary heathy adults
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Sway Velocity | April 2021 - May 2021
  the average displacement of CoP per second
Sway area | April 2021 - May 2021
  total area obtained by the displacement of the COP
Perimeter | April 2021 - May 2021
  the total displacement of CoP

CONTACTS AND LOCATIONS:
Overall Officials: Sahra Şirvan Can, Master's, Principal Investigator — Yeditepe University; Çiğdem v, PhD, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asslander L, Streuber S. Virtual reality as a tool for balance research: Eyes open body sway is reproduced in photo-realistic, but not in abstract virtual scenes. PLoS One. 2020 Oct 29;15(10):e0241479. doi: 10.1371/journal.pone.0241479. eCollection 2020. PMID 33119679
- [Result] Chander H, Kodithuwakku Arachchige SNK, Hill CM, Turner AJ, Deb S, Shojaei A, Hudson C, Knight AC, Carruth DW. Virtual-Reality-Induced Visual Perturbations Impact Postural Control System Behavior. Behav Sci (Basel). 2019 Nov 12;9(11):113. doi: 10.3390/bs9110113. PMID 31718105